CLINICAL TRIAL: NCT03087188
Title: Inhalation Therapy in Ambulant and Hospitalized Patient Using Available Film Sequences From the Internet
Acronym: InhaliPAD
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 15-031
Record Dates: First submitted 2017-03-15; First posted 2017-03-22 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Obstructive Lung Disease; COPD; Asthma
MeSH Terms: conditions — Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Utilization of inhalator: Film sequences will be shown to patients using incorrect application technique in order to improve technique. Learning success will be assessed subsequently and at a follow-up visit after 2-8 weeks
  Interventions: Other: Utilization of inhalator

INTERVENTIONS:
Other: Utilization of inhalator — After written consent patients will be asked whether they know how to use the inhalator and for how long therapy has been already conducted. Patients using the inhalator correctly have completed the study at this point. If patients have demonstrated incorrect use of the inhalator, a film sequence with instructions will be shown via a tablet. The learning success will be assessed subsequently. When patients show correct application, they will be asked to come back for a follow-up visit within 2 to 8 weeks, otherwise they will be retrained by study staff. At the follow-up visit another demonstration evaluation will be performed.
  While demonstrating patients will use the inhalator without any drug that could have any medicinal effect on them.

SUMMARY:
There are different therapy strategies for patients suffering on obstructive lung disease like chronic obstructive pulmonary disease (COPD), and asthma bronchial available. One of these strategies includes inhalative drugs, e.g. ß2-mimetics, anticholinergic drugs, or glucocorticoids, which are indicated often and which can be used with different inhalation devices. Dry powder inhalators, and dosieraerosol are used the most in clinical routine. Further strategies in treating obstructive lung disease are innovative systems like Respimat or systems with liquid inhalation. However, the success of the therapy depends on the correct application technique. In the clinical routine a high error rate was observed. Consequently, the initiative of the German league of respiratory tracts published internet-based film sequences in order to demonstrate how to use an inhalator correctly. These films are available in the internet for everyone and can be watched as often as needed in order to improve technique and facilitate training.

Therefore, in this study we aim to evaluate the following aspects:

* amount of wrong applications in ambulant and hospitalized patients (wrong in terms of lack of knowledge on how to use the inhalator or incorrect utilization)
* amount of correct applications in patients who had first used the inhalator incorrectly but improved technique by watching the film sequences
* evaluation of learning success within 2 weeks to 2 months (follow-up visit in the ambulance)

ELIGIBILITY:
Inclusion Criteria:

* male and female patients indicated for inhalative treatment with ß2-mimetics, inhalative steroids, anticholinergic drugs, or a combination of these drugs
* patient was already trained on how to use the inhalator before participating in the study
* age > 18
* obtained written consent

Exclusion Criteria:

* patients who are incapable to consent or are unable to understand the scope of the trial
* patients who indicate that they do not know how to use the inhalator

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients in need of inhalative therapy due to obstructive lung disease, COPD, or asthma bronchial
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2015-09-09 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Correct utilization of inhalator | Day of Screening and follow-up visit (2-8 weeks)
  Wrong utilization is determined as lack of knowledge on how to use the inhalator or incorrect application

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Müller, PD Dr. med., Principal Investigator — University Hospital, Aachen
Locations (1):
- University Hospital RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided